CLINICAL TRIAL: NCT00278850
Title: "Vestibulitis Educational Seminar Trial" Study
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Lori Brotto, Associate Professor, University of British Columbia
Other Study IDs: C05-0592
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Vulvar Vestibulitis
Keywords: Vulvar vestibulitis; Treatment; Education
MeSH Terms: conditions — Vulvar Vestibulitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Educational — three 1 hour long educational seminars

SUMMARY:
The purpose of this study is to investigate the efficacy of an educational seminar series for women with vulvar vestibulitis syndrome (VVS).

DETAILED DESCRIPTION:
HYPOTHESIS: It is hypothesized that this educational seminar series might be effective in reducing the pain experienced and improving sexual response and quality of life of women with Vulvar Vestibulitis Syndrome (VVS) by providing an open forum for discussion of the pathology, etiological theories, treatment plans as well as the impact of sexual pain on sexual relationships and ways to cope with VVS.

At Vancouver Hospital, the current waitlist for women with distressing, unremitting genital pain is approximately 10 months. Once accepted for management, the diagnosis of VVS is given, where applicable, by Dr. Sadownik. Only women with pure VVS and without a compounding skin condition are then referred on to the 3-session educational seminars given by Dr. Thomson. By the end of the educational series, women have an understanding of current scientific literature on etiology and treatment of VVS, and it's interaction with sexual health factors. At this point they are referred for individualized treatment of the VVS either by Dr. Thomson, Dr. Sadownik or back to their referring physician. This study aims to explore the existing VVS Educational Seminars by measuring sexual function, sexual distress, pain levels (general pain, genital pain and pain upon sexual activity), psychological well-being (depression and anxiety), relationship satisfaction, sexual knowledge and overall quality of life at pre- and post seminar. An age-matched control group of women diagnosed with VVS, but unable to attend the Seminar series, will complete the measures at the same intervals as the treatment group. The use of the control group allows us to accurately evaluate the efficacy of the Educational seminars, above and beyond non-specific factors.

Vulvar Vestibulitis Syndrome Educational Seminars have been run through the Vulvar Disease Clinic at Vancouver Hospital since 2001, however no data has been collected to determine the effects of this program. By collecting pre- & post seminar and follow up data, this study will allow us to assess the efficacy of the VVS Educational Seminars when compared to a group of women suffering from VVS but unable to attend the information seminars. Given that a large proportion of the women cannot be treated at Vancouver Hospital and are instead referred back to their family physician, the VVS Educational Seminar is a necessary first step in the treatment process for ensuring that women receive accurate and timely treatment. It will also help treatment providers improve and expand their current treatment practices

ELIGIBILITY:
Inclusion Criteria:

* Women who meet the diagnostic criteria for VVS by the Vancouver Hospital Vulvar Disease Clinic
* Women who have been referred to VVS Educational Seminars at Vancouver Hospital
* Proficient in English

Exclusion Criteria:

* Any women referred to the VVS Educational Seminars will be eligible for participation.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women diagnosed with vulvar vestibulitis
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2006-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori A Brotto, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Abramov L, Wolman I, David MP. Vaginismus: an important factor in the evaluation and management of vulvar vestibulitis syndrome. Gynecol Obstet Invest. 1994;38(3):194-7. doi: 10.1159/000292478. PMID 8001875
- [Background] Bergeron S, Binik YM, Khalife S, Pagidas K, Glazer HI. Vulvar vestibulitis syndrome: reliability of diagnosis and evaluation of current diagnostic criteria. Obstet Gynecol. 2001 Jul;98(1):45-51. doi: 10.1016/s0029-7844(01)01389-8. PMID 11430955
- [Background] Bergeron S, Binik YM, Khalife S, Pagidas K. Vulvar vestibulitis syndrome: a critical review. Clin J Pain. 1997 Mar;13(1):27-42. doi: 10.1097/00002508-199703000-00006. PMID 9084950
- [Background] Bornstein J, Livnat G, Stolar Z, Abramovici H. Pure versus complicated vulvar vestibulitis: a randomized trial of fluconazole treatment. Gynecol Obstet Invest. 2000;50(3):194-7. doi: 10.1159/000010309. PMID 11014954
- [Background] Pukall CF, Payne KA, Binik YM, Khalife S. Pain measurement in vulvodynia. J Sex Marital Ther. 2003;29 Suppl 1:111-20. doi: 10.1080/713847136. PMID 12735095
- [Background] Bergeron, S., Binik, YM., Khalifé, S., Meana, M., Berkely, KJ. & Pagidas, K. (1997). The treatment of vulvar vestibulitis syndrome: Towards a multimodal approach. Sexual & Marital Therapy, 12(4), 305-311.
- [Background] Glazer HI, Rodke G, Swencionis C, Hertz R, Young AW. Treatment of vulvar vestibulitis syndrome with electromyographic biofeedback of pelvic floor musculature. J Reprod Med. 1995 Apr;40(4):283-90. PMID 7623358
- [Background] Pukall, C.F., Payne, K.A., Kao, A., Khalife, S. & Binik, Y.M. (2005). Dyspareunia. In R. Balon & R.T. Segraves, (Ed.s), Handbook of Sexual Dysfunction (pp. 249-272). New York: Taylor and Francis.
- [Background] ter Kuile, MM. & Weijenborg, ThM, (2003). A cognitive behavioural group treatment programme for women with vulvar vestibulitis syndrome: factors associated with treatment success. Sexual Pain Disorders Symposium, Amsterdam, Holland, Oct. 20-24, 2003.
- [Background] Friedrich EG Jr. Vulvar vestibulitis syndrome. J Reprod Med. 1987 Feb;32(2):110-4. PMID 3560069
- [Background] Schover LR, Youngs DD, Cannata R. Psychosexual aspects of the evaluation and management of vulvar vestibulitis. Am J Obstet Gynecol. 1992 Sep;167(3):630-6. doi: 10.1016/s0002-9378(11)91562-2. PMID 1530015
- [Background] Weijmar Schultz WC, Gianotten WL, van der Meijden WI, van de Wiel HB, Blindeman L, Chadha S, Drogendijk AC. Behavioral approach with or without surgical intervention to the vulvar vestibulitis syndrome: a prospective randomized and non-randomized study. J Psychosom Obstet Gynaecol. 1996 Sep;17(3):143-8. doi: 10.3109/01674829609025675. PMID 8892160